CLINICAL TRIAL: NCT03772535
Title: Using Pharmacogenetics to Structure Individual Pain Management Protocols for Joint Replacement Patients
Brief Title: Pharmacogenetics for Pain Management in Joint Replacement Patients
Acronym: PGx
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Anderson Orthopaedic Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: AORI 2018-0100
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Arthroplasty Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (No Intervention): Subjects in this arm will receive the standard postoperative pain prescription protocol.
- Pharmacogenomics Guided Group (Active Comparator): Subjects in this group will receive postoperative pain prescriptions based on the results of pharmacogenomic testing.
  Interventions: Diagnostic Test: Pharmacogenomics Testing

INTERVENTIONS:
Diagnostic Test: Pharmacogenomics Testing — The doctor will use genetic test results to prescribe medications that are a most effective for subject.
  Arms: Pharmacogenomics Guided Group

SUMMARY:
The purpose of this study is to determine the ability to use pharmacogenetic testing in a joint replacement practice to prescribe the most effective pain medicine for a specific patient.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip or total knee arthroplasty cases

Exclusion Criteria:

* History of narcotic dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variants | 10 days postoperative
  Percent of subject with genetic variants affecting pain medication

SECONDARY OUTCOMES:
pain levels | 10 days postoperatively
  0-10 subjective pain scale

CONTACTS AND LOCATIONS:
Overall Officials: William Hamilton, MD, Principal Investigator — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States